CLINICAL TRIAL: NCT06708117
Title: Exploring the Effects of Obesity and Bariatric Surgery on the Brain Using Magnetic Resonance Imaging
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202406090RINA
Record Dates: First submitted 2024-11-19; First posted 2024-11-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: obesity; bariatric surgery; brain; magnetic resonance imaging
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background and Purpose:

The causes of obesity are highly complex, with eating behaviors playing a crucial role. Current research indicates that many brain regions are involved in the regulation of appetite, eating behaviors, and obesity, but the detailed mechanisms remain unclear. Bariatric surgery has been shown to effectively achieve long-term weight loss and improve obesity-related conditions in severely obese patients, making it a valuable research platform for obesity treatment. Recent studies have found that after bariatric surgery, patients experience reduced hunger, increased satiety, and altered responses and preferences for food stimuli. Magnetic resonance imaging (MRI) is a widely used tool for analyzing brain structure and functional changes. Recent imaging studies have demonstrated changes in brain structure and connectivity across multiple regions after bariatric surgery. However, due to the complexity of brain structure and these changes, many questions remain unanswered. This study aims to investigate the effects of obesity and bariatric surgery on brain structure and function using MRI, to identify potential mechanisms for treating obesity.

Methods:

This study plans to recruit 200 obese patients aged 20 years or older who are scheduled to undergo bariatric surgery within a 5-year period. Participants will undergo brain MRI scans before and six months after surgery. At these two time points, they will also complete the Dutch Eating Behavior Questionnaire (DEBQ) to assess changes in eating behaviors and provide blood samples for the analysis of gastrointestinal, obesity-related, and appetite-related hormones. Additionally, 60 healthy individuals with normal weight will be recruited as a control group to undergo the same brain MRI scans, DEBQ assessments, and blood analyses. This control group will help explore the effects of obesity and bariatric surgery on brain structure and function.

Expected Results:

This study is expected to reveal the structural and functional changes in brain MRI associated with obesity and bariatric surgery, providing insights into potential mechanisms for treating obesity.

DETAILED DESCRIPTION:
A. Bariatric Surgery Participants Obese patients scheduled for bariatric surgery will be recruited through the Bariatric Surgery Outpatient Clinic of the Department of Surgery at National Taiwan University Hospital (NTUH). Physicians and research staff will explain the study procedures to the patients.

B. Healthy Normal-Weight Participants Healthy participants will be recruited via promotional materials distributed within NTUH and online. Physicians and research staff will explain the study procedures to the participants.

ELIGIBILITY:
A. Bariatric Surgery Participants

Inclusion Criteria (Eligibility for Study Participation):

* Aged 20 years or older.
* Body mass index (BMI) ≥ 37.5, or BMI ≥ 27 with obesity-related comorbidities such as type 2 diabetes, hypertension, or obstructive sleep apnea.
* Scheduled to undergo bariatric surgery for obesity treatment.

Exclusion Criteria:

* Presence of neurological or psychiatric disorders.
* Use of neurological or psychiatric medications.
* Diagnosis of cancer or major gastrointestinal diseases.
* History of major abdominal surgery.
* Presence of metallic implants in the body.
* Claustrophobia.
* Currently pregnant.

B. Healthy Normal-Weight Participants

Inclusion Criteria (Eligibility for Study Participation):

* Aged 20 to 65 years.
* BMI between 18.5 and 24.

Exclusion Criteria:

* Presence of neurological or psychiatric disorders.
* Use of neurological or psychiatric medications.
* Diagnosis of cancer or major gastrointestinal diseases.
* History of major abdominal surgery.
* Presence of metallic implants in the body.
* Claustrophobia.
* Currently pregnant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A. Bariatric Surgery Participants B. Healthy Normal-Weight Participants
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Bariatric surgery-related structural changes as assessed by gray matter volume | Baseline and 6 months after bariatric surgery
  Acquiring structural brain MR images before and six months after bariatric surgery
Bariatric surgery-related changes in functional connection between brain areas as assessed by Pearson's correlation coefficient | Baseline and 6 months after bariatric surgery
  Performing resting-state functional MRI before and six months after bariatric surgery
Obesity-related structural changes as assessed by gray matter volume | From enrollment to brain MRI
  Acquiring structural brain MR images in health controls and bariatric patents before surgery
Obesity-related changes in functional connection between brain areas as assessed by Pearson's correlation coefficient | From enrollment to brain MRI
  Performing resting-state functional MRI in health controls and bariatric patents before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Po-Jen Yang, MD, PhD, Principal Investigator — National Taiwan University Hospital